CLINICAL TRIAL: NCT05924321
Title: A Randomized, 2-Part, Crossover Trial to Evaluate the Effect of Carbetocin on the QT/QTc Interval in Healthy Subjects
Brief Title: A Study to Evaluate the Effect of Carbetocin on the QT/QTc Interval in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 000421
Record Dates: First submitted 2023-05-03; First posted 2023-06-29 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2023-05

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — carbetocin; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The trial will consist of two parts; Part A and Part B. Part A is an open-label single group trial while Part B is a double-blind trial with 3 groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Carbetocin (Experimental): Single IV infusion of carbetocin
  Interventions: Drug: Carbetocin
- Placebo (Placebo Comparator): Single IV Infusion of matching placebo
  Interventions: Drug: Placebo
- Placebo and Moxifloxacin (Active Comparator): Single IV infusion of matching placebo with a single oral dose of moxifloxacin
  Interventions: Drug: Placebo and Moxifloxacin

INTERVENTIONS:
Drug: Carbetocin — Single infusion of Carbetocin
  Arms: Carbetocin
Drug: Placebo — Single IV infusion of matching placebo
  Arms: Placebo
Drug: Placebo and Moxifloxacin — Single IV infusion of matching placebo in combination with Single Oral dose of Moxifloxacin
  Arms: Placebo and Moxifloxacin

SUMMARY:
Carbetocin is an oxytocin receptor agonist that selectively binds to receptors in the smooth muscle of the uterus, stimulates rhythmic contractions of the uterus, increases the frequency of existing contractions, and raises the tone of the uterine musculature. Carbetocin is approved in >100 countries for the prevention of postpartum hemorrhage due to uterine atony in women following cesarean or vaginal delivery. Per regulatory requirements, the current trial will evaluate the effects of high clinical exposure of carbetocin on the QT interval corrected for heart rate (QTc) as measured by ECG in healthy men and women.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, male or female subjects, 18-45 years of age, inclusive, at the screening visit.
* Body mass index (BMI) ≥ 18.5 and ≤29.9 kg/m2 at the screening visit.
* Continuous non-smoker who has not used nicotine- or tobacco-containing products for at least 3 months prior to first dosing.

Exclusion Criteria:

* Sustained supine systolic blood pressure ≥130 mmHg or <90 mmHg, supine diastolic blood pressure ≥80 mmHg or <50 mmHg at screening or first check-in.
* History or presence of clinically significant ECG findings in the opinion of the Principal Investigator (PI) or designee at the screening visit or first check-in, including each of the following:

  * HR <45 bpm or >100 bpm.
  * QTcF is ≥450 msec (males) or ≥460 msec (females).
  * QRS ≥110 msec; if ≥110 msec, result will be confirmed by a manual over read.
  * PR ≥200 msec.
* History or presence of:

  * Risk factors for Torsades de Pointes (e.g., heart failure, cardiomyopathy, family history of Long QT syndrome, Brugada syndrome, or sudden cardiac death).
  * Sick sinus syndrome, second- or third-degree atrioventricular block, myocardial infarction, angina, pulmonary congestion, symptomatic or significant cardiac arrhythmia, or clinically significant conduction abnormalities.
  * Clinically significant abnormal laboratory assessments including hypokalemia, hypercalcemia, or hypomagnesemia, in the opinion of the PI or designee.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-09-21 (Actual)

PRIMARY OUTCOMES:
Observed Heart rate(HR) values | Up to 240 minutes after Start of Infusion
  Part A
Change from baseline of HR (∆HR). | Up to 240 minutes after Start of Infusion
  Part A
Placebo-corrected change from baseline in QT interval (∆∆QTc) using the most appropriate HR correction method (i.e., ∆∆QTcF if Fridericia's method is used). | Up to 24 hours after Start of Infusion
  Part B

SECONDARY OUTCOMES:
Treatment-emergent adverse events (TEAEs) | Up to follow-up visit (7 to 10 days after the last dose)
  Part A
Vital signs; Systolic blood pressure and Diastolic blood pressure | Up to follow-up visit (7 to 10 days after the last dose)
  Part A. The parameters which are measured are Systolic blood pressure and Diastolic blood pressure.
  Each vital sign parameter value is classified as either Low, Normal or High. Summary tables will be prepared by treatment displaying the number and percentage of subjects with normal pre-administration values who had at least one markedly abnormal post-administration values.
Vital signs; Pulse rate | Up to follow-up visit (7 to 10 days after the last dose)
  Part A. The parameter which is measured is Pulse rate. The vital sign parameter value is classified as either Low, Normal or High. Summary tables will be prepared by treatment displaying the number and percentage of subjects with normal pre-administration values who had at least one markedly abnormal post-administration values.
Vital signs; Body temperature | Up to follow-up visit (7 to 10 days after the last dose)
  Part A. The parameter which is measured is Body temperature. The vital sign parameter value is classified as either Low, Normal or High. Summary tables will be prepared by treatment displaying the number and percentage of subjects with normal pre-administration values who had at least one markedly abnormal post-administration values.
Vital signs; Respiratory rate | Up to follow-up visit (7 to 10 days after the last dose)
  Part A. The parameter which is measured is Respiratory rate. The vital sign parameter value is classified as either Low, Normal or High. Summary tables will be prepared by treatment displaying the number and percentage of subjects with normal pre-administration values who had at least one markedly abnormal post-administration values.
12-lead safety ECGs | Up to follow-up visit (7 to 10 days after the last dose)
  Part A. The parameters which are measured are QT, QTc, QTcF, QRS, PR, RR and HR. Subjects' maximum change from baseline and subject's maximum post-baseline values in ECG parameters will be categorized and the number and percentage of subjects in each group will be summarized.
  The results will be interpreted as "normal", "abnormal, not clinically significant" or "abnormal clinically significant", and the interpretation will be summarized for each treatment and scheduled time point using frequency counts and percentages.
Clinical chemistry: Changes in Concentration of Blood Urea Nitrogen | Up to follow-up visit (7 to 10 days after the last dose)
  Part A. Assessed by blood sample collection
Clinical chemistry: Changes in Concentration of Bilirubin Total | Up to follow-up visit (7 to 10 days after the last dose)
  Part A. Assessed by blood sample collection
Clinical chemistry: Changes in Concentration of Bilirubin direct | Up to follow-up visit (7 to 10 days after the last dose)
  Part A. Assessed by blood sample collection
Clinical chemistry: Changes in Concentration of Alkaline phosphatase | Up to follow-up visit (7 to 10 days after the last dose)
  Part A. Assessed by blood sample collection
Clinical chemistry: Changes in Concentration of Aspartate aminotransferase | Up to follow-up visit (7 to 10 days after the last dose)
  Part A. Assessed by blood sample collection
Clinical chemistry: Changes in Concentration of Alanine aminotransferase | Up to follow-up visit (7 to 10 days after the last dose)
  Part A. Assessed by blood sample collection
Clinical chemistry: Changes in Concentration of Albumin | Up to follow-up visit (7 to 10 days after the last dose)
  Part A. Assessed by blood sample collection
Clinical chemistry: Changes in Concentration of Sodium | Up to follow-up visit (7 to 10 days after the last dose)
  Part A. Assessed by blood sample collection
Clinical chemistry: Changes in Concentration of Potassium | Up to follow-up visit (7 to 10 days after the last dose)
  Part A. Assessed by blood sample collection
Clinical chemistry: Changes in Concentration of Magnesium | Up to follow-up visit (7 to 10 days after the last dose)
  Part A. Assessed by blood sample collection
Clinical chemistry: Changes in Concentration of Chloride | Up to follow-up visit (7 to 10 days after the last dose)
  Part A. Assessed by blood sample collection
Clinical chemistry: Changes in Concentration of Fasting glucose | Up to follow-up visit (7 to 10 days after the last dose)
  Part A. Assessed by blood sample collection
Clinical chemistry: Changes in Concentration of Creatinine | Up to follow-up visit (7 to 10 days after the last dose)
  Part A. Assessed by blood sample collection
Hematology: Changes in Concentration of Hemoglobin | Up to follow-up visit (7 to 10 days after the last dose)
  Part A. Assessed by blood sample collection
Hematology: Changes in Concentration of Hematocrit | Up to follow-up visit (7 to 10 days after the last dose)
  Part A. Assessed by blood sample collection
Hematology: Changes in Concentration of Total and differential leukocyte count | Up to follow-up visit (7 to 10 days after the last dose)
  Part A. Assessed by blood sample collection
Hematology: Changes in Concentration of Red blood cell count | Up to follow-up visit (7 to 10 days after the last dose)
  Part A. Assessed by blood sample collection
Hematology: Changes in Concentration of Platelet count | Up to follow-up visit (7 to 10 days after the last dose)
  Part A. Assessed by blood sample collection
Urinalysis parameters: Concentration of pH | Up to follow-up visit (7 to 10 days after the last dose)
  Part A. Assessed by urine sample collection
Urinalysis parameters: Concentration of specific gravity | Up to follow-up visit (7 to 10 days after the last dose)
  Part A. Assessed by urine sample collection
Urinalysis parameters: Concentration of Protein | Up to follow-up visit (7 to 10 days after the last dose)
  Part A. Assessed by urine sample collection
Urinalysis parameters: Concentration of Glucose | Up to follow-up visit (7 to 10 days after the last dose)
  Part A. Assessed by urine sample collection
Urinalysis parameters: Concentration of Bilirubin | Up to follow-up visit (7 to 10 days after the last dose)
  Part A. Assessed by urine sample collection
Urinalysis parameters: Concentration of Blood | Up to follow-up visit (7 to 10 days after the last dose)
  Part A. Assessed by urine sample collection
Urinalysis parameters: Concentration of Nitrite | Up to follow-up visit (7 to 10 days after the last dose)
  Part A. Assessed by urine sample collection
Urinalysis parameters: Concentration of Urobilinogen | Up to follow-up visit (7 to 10 days after the last dose)
  Part A. Assessed by urine sample collection
Urinalysis parameters: Concentration of Leukocyte esterase | Up to follow-up visit (7 to 10 days after the last dose)
  Part A. Assessed by urine sample collection
∆HR, PR change from baseline (∆PR), RR change from baseline (∆RR), QRS change from baseline (∆QRS), and QTcF change from baseline (∆QTcF), if not selected as the primary endpoint. | Up to 24 hours after Start of Infusion
  Part B
Placebo-corrected ∆HR (∆∆HR), placebo-corrected ∆PR (∆∆PR), placebo-corrected ∆RR (∆∆RR), placebo-corrected ∆QRS (∆∆QRS), and ∆∆QTcF, if not selected as the primary endpoint | Up to 24 hours after Start of Infusion
  Part B
Categorical outliers for QTcF | Up to 24 hours after Start of Infusion
  Part B
Categorical outliers for HR | Up to 24 hours after Start of Infusion
  Part B
Categorical outliers for PR | Up to 24 hours after Start of Infusion
  Part B
Categorical outliers for QRS | Up to 24 hours after Start of Infusion
  Part B
Abnormalities in T wave morphology and pathologic U waves, as appropriate. | Up to 24 hours after Start of Infusion
  Part B
Carbetocin PK parameters: AUClast | Up to 24 hours after Start of Infusion
  Part B
Carbetocin PK parameters: AUCinf | Up to 24 hours after Start of Infusion
  Part B
Carbetocin PK parameters: AUC%extrap | Up to 24 hours after Start of Infusion
  Part B
Carbetocin PK parameters: Cmax | Up to 24 hours after Start of Infusion
  Part B
Carbetocin PK parameters: Tmax | Up to 24 hours after Start of Infusion
  Part B
Carbetocin PK parameters: t½ | Up to 24 hours after Start of Infusion
  Part B
Carbetocin PK parameters: MRTinf | Up to 24 hours after Start of Infusion
  Part B
Carbetocin PK parameters: CL | Up to 24 hours after Start of Infusion
  Part B
Carbetocin PK parameters: Vss | Up to 24 hours after Start of Infusion
  Part B
Carbetocin PK parameters: Vz. | Up to 24 hours after Start of Infusion
  Part B
∆∆QTc (i.e., ∆∆QTcF or the most appropriate HR correction method) following administration of moxifloxacin. | Up to 24 hours after Start of Infusion
  Part B
TEAEs | End of Trial (Up to 25 days)
  Part B
Vital signs; Systolic blood pressure and Diastolic blood pressure | End of Trial (Up to 25 days)
  Part B. The parameters which are measured are Systolic blood pressure and Diastolic blood pressure.
  Each vital sign parameter value is classified as either Low, Normal or High
Vital signs; Pulse rate | End of Trial (Up to 25 days)
  Part B. The parameter which is measured is Pulse rate. The sign parameter value is classified as either Low, Normal or High
Vital signs; Body temperature | End of Trial (Up to 25 days)
  Part B. The parameter which is measured is Body temperature. The sign parameter value is classified as either Low, Normal or High
Vital signs; Respiratory rate | End of Trial (Up to 25 days)
  Part B. The parameter which is measured is Respiratory rate. The sign parameter value is classified as either Low, Normal or High
12-lead safety ECGs | End of Trial (Up to 25 days)
  Part B. The parameters which are measured are QT, QTc, QTcF, QRS, PR, RR and HR. The results will be interpreted as "normal", "abnormal, not clinically significant" or "abnormal clinically significant".
Clinical chemistry: Changes in Concentration of Blood Urea Nitrogen | End of Trial (Up to 25 days)
  Part B. Assessed by blood sample collection
Clinical chemistry: Changes in Concentration of Bilirubin total | End of Trial (Up to 25 days)
  Part B. Assessed by blood sample collection
Clinical chemistry: Changes in Concentration of Bilirubin direct | End of Trial (Up to 25 days)
  Part B. Assessed by blood sample collection
Clinical chemistry: Changes in Concentration of Alkaline phosphatase | End of Trial (Up to 25 days)
  Part B. Assessed by blood sample collection
Clinical chemistry: Changes in Concentration of Aspartate aminotransferase | End of Trial (Up to 25 days)
  Part B. Assessed by blood sample collection
Clinical chemistry: Changes in Concentration of Alanine aminotransferase | End of Trial (Up to 25 days)
  Part B. Assessed by blood sample collection
Clinical chemistry: Changes in Concentration of Albumin | End of Trial (Up to 25 days)
  Part B. Assessed by blood sample collection
Clinical chemistry: Changes in Concentration of Sodium | End of Trial (Up to 25 days)
  Part B. Assessed by blood sample collection
Clinical chemistry: Changes in Concentration of Potassium | End of Trial (Up to 25 days)
  Part B. Assessed by blood sample collection
Clinical chemistry: Changes in Concentration of Magnesium | End of Trial (Up to 25 days)
  Part B. Assessed by blood sample collection
Clinical chemistry: Changes in Concentration of Chloride | End of Trial (Up to 25 days)
  Part B. Assessed by blood sample collection
Clinical chemistry: Changes in Concentration of Fasting glucose | End of Trial (Up to 25 days)
  Part B. Assessed by blood sample collection
Clinical chemistry: Changes in Concentration of Creatinine | End of Trial (Up to 25 days)
  Part B. Assessed by blood sample collection
Hematology: Changes in Concentration of Hemoglobin | End of Trial (Up to 25 days)
  Part B. Assessed by blood sample collection
Hematology: Changes in Concentration of Hematocrit | End of Trial (Up to 25 days)
  Part B. Assessed by blood sample collection
Hematology: Changes in Concentration of Total and Differential leukocyte count | End of Trial (Up to 25 days)
  Part B. Assessed by blood sample collection
Hematology: Changes in Concentration of Red blood cell count | End of Trial (Up to 25 days)
  Part B. Assessed by blood sample collection
Hematology: Changes in Concentration of Platelet count | End of Trial (Up to 25 days)
  Part B. Assessed by blood sample collection
Urinalysis parameters: Concentration of pH | End of Trial (Up to 25 days)
  Part B. Assessed by urine sample collection
Urinalysis parameters: Concentration of Specific gravity | End of Trial (Up to 25 days)
  Part B. Assessed by urine sample collection
Urinalysis parameters: Concentration of Protein | End of Trial (Up to 25 days)
  Part B. Assessed by urine sample collection
Urinalysis parameters: Concentration of Glucose | End of Trial (Up to 25 days)
  Part B. Assessed by urine sample collection
Urinalysis parameters: Concentration of Bilirubin | End of Trial (Up to 25 days)
  Part B. Assessed by urine sample collection
Urinalysis parameters: Concentration of Blood | End of Trial (Up to 25 days)
  Part B. Assessed by urine sample collection
Urinalysis parameters: Concentration of Nitrite | End of Trial (Up to 25 days)
  Part B. Assessed by urine sample collection
Urinalysis parameters: Concentration of Urobilinogen | End of Trial (Up to 25 days)
  Part B. Assessed by urine sample collection
Urinalysis parameters: Concentration of Leukocyte esterase | End of Trial (Up to 25 days)
  Part B. Assessed by urine sample collection

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (1):
- Ferring Investigational Site, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No